CLINICAL TRIAL: NCT01982578
Title: Effect of Activation of the Receptor PPARg/RXR as a Possible Treatment for Alzheimer's Disease. Role of Genistein.
Brief Title: Genistein as a Possible Treatment for Alzheimer's Disease.
Acronym: GENIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Collaborators: University of Valencia (Other)
Responsible Party: Principal Investigator, Jose Vina, Professor M.D. Ph. D. (hon), Fundación para la Investigación del Hospital Clínico de Valencia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INC-GEN-2013-01; U1111-1150-4063 (Other: World Health Organization)
Record Dates: First submitted 2013-10-30; First posted 2013-11-13 (Estimated); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Alzheimer's Disease
Keywords: Treatment; Genistein; Alzheimer's disease; Cerebrospinal fluid; Amyloid beta
MeSH Terms: conditions — Alzheimer Disease; Plaque, Amyloid | interventions — Genistein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Product: Genistein (Experimental): 60 mg of genistein BID for 360 days. Intervention: Product: Genistein
  Interventions: Dietary Supplement: Genistein
- Product: Placebo (Placebo Comparator): 1 placebo capsule BID for 360 days. Intervention: Product: Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Genistein — Subjects will be randomized 1:1 to receive 360 days of double blind treatment of genistein.
  Other Names: Fisiogen
  Arms: Product: Genistein
Other: Placebo — 360 days of double blind treatment of placebo.
  Arms: Product: Placebo

SUMMARY:
Genistein is an isoflavone that has antioxidant and neuroprotective effects on Alzheimer's disease (AD).

A few years ago our group reported that genistein increased PPARg (peroxisome proliferator activated receptor gamma) levels. By the way, activation of retinoid X receptor (RXR)-PPARg dimer, will make overexpressing apolipoprotein E (apoE), which mediates the degradation of amyloid beta (AB). Therefore, we believe that if this phytoestrogen administration increases the availability of the transcription factor, it can increase apoE, and also AB degradation.

The main aim of this study is to determinate the effect of 60 mg BID of genistein administration, during 360 days, compared to placebo group, in AD patients.

DETAILED DESCRIPTION:
Alzheimer's disease is devastating in terms of personal wellbeing as well as for society. Any effort to prevent and/or treat this disease is always sought after. Recently, an exciting new possibility was opened by modulating a cellular component called RXR-PPARG. A successful experimental treatment for Alzheimer's was found by activating RXR. But we previously showed that a component of soya, i.e., genistein, is able to activate the other part of the RXR-PPARG molecule, i.e., the PPARG moiety. Genistein, moreover, does not have the undesirable effect of bexarotene and is a food component. Our preliminary results in animals indicate that genistein is effective in the treatment of experimental Alzheimer's in mice. Epidemiological evidence shows that individuals who live in Eastern societies who have a high genistein intake (because they eat a lot of soya) have lower rates of Alzheimer's disease.

Thus we propose a controlled clinical trial to test if administration of the food component genistein is able to prevent or cure, at least partially, Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild cognitive impairment (MCI) compatible with prodromal AD.
* Mini-Mental State Examinations (MMSE) score between over 24 inclusive.
* CSF levels of AB, p-TAU compatible with AD.
* 18 years or older.
* Must have a study partner who is able and willing to comply with all required study procedures.
* Willing and able to provide informed consent by either the subject or subject's legal representative.

Exclusion Criteria:

* Patient who does not meet the inclusion criteria.
* Thyroid abnormalities with or without treatment.
* Immune abnormalities in blood analyses.
* Patient suffers hormone dependent neoplasia.
* Take a diet rich on isoflavones.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in Amyloid beta concentration in cerebrospinal fluid (CSF) | Day 0 and day 360 (plus or minus 7 day)
  The primary study endpoint is the change from baseline to the end of the treatment, and the change between the treatment group and the placebo group.

SECONDARY OUTCOMES:
Changes in MMSE. | Day 0, day 180, day 360, (plus or minus 7 days)
  Change from baseline to the end of the treatment, and the change between the treatment group and the placebo group.
Changes in T@M (Memory Alteration Test). | Day 0, day 180, day 360, (plus or minus 7 days)
  Change from baseline to the end of the treatment, and the change between the treatment group and the placebo group.This is a memory screening test, capable for discriminating between subjects with subjective memory complaints (SMC) (without objective memory impairment) and patients with amnestic mild cognitive impairment (A-MCI) and with mild Alzheimer's disease (AD) (Archives of Gerontology and Geriatrics. 2010 Mar-Apr;50(2):171-4. doi: 10.1016/j.archger.2009.03.005. Epub 2009 Apr 16)
Changes in TAVEC (Verbal Learning Test Spain-COmplutense). | Day 0, day 180, day 360, (plus or minus 7 days)
  Change from baseline to the end of the treatment, and the change between the treatment group and the placebo group.
Changes in the Clock test. | Day 0, day 180, day 360, (plus or minus 7 days)
  Change from baseline to the end of the treatment, and the change between the treatment group and the placebo group.
Changes in the Barcelona Test. | Day 0, day 180, day 360, (plus or minus 7 days)
  Change from baseline to the end of the treatment, and the change between the treatment group and the placebo group.
Changes in Rey Complex figure Test. | Day 0, day 180, day 360, (plus or minus 7 days)
  Change from baseline to the end of the treatment, and the change between the treatment group and the placebo group.
Changes in Genistein Pharmacokinetics. | Day 0, day 360, (plus or minus 7 days)
  Change from baseline to the end of the treatment,and the change between the treatment group and the placebo group.
Changes in Equol Pharmacokinetics. | Day 0, day 360, (plus or minus 7 days)
  Change from baseline to the end of the treatment,and the change between the treatment group and the placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Viña, MD PhD (hon), Principal Investigator — University of Valencia
Locations (2):
- Spain (2):
  - Universitat de València, Valencia
  - Hospital General Universitario, Valencia

REFERENCES:
- [Derived] Vina J, Escudero J, Baquero M, Cebrian M, Carbonell-Asins JA, Munoz JE, Satorres E, Melendez JC, Ferrer-Rebolleda J, Cozar-Santiago MDP, Santabarbara-Gomez JM, Jove M, Pamplona R, Tarazona-Santabalbina FJ, Borras C. Genistein effect on cognition in prodromal Alzheimer's disease patients. The GENIAL clinical trial. Alzheimers Res Ther. 2022 Nov 4;14(1):164. doi: 10.1186/s13195-022-01097-2. PMID 36329553